CLINICAL TRIAL: NCT03148808
Title: Natural Vascular Scaffold (NVS) Therapy for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA)
Brief Title: Natural Vascular Scaffold (NVS) Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alucent Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol No.: 1060-001
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases; Catheterization, Peripheral
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: NVS Therapy will be delivered to de novo lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) during PTA in patients with symptomatic peripheral artery disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NVS Therapy (Experimental): NVS Therapy will be delivered to de novo lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) during PTA in patients with symptomatic peripheral artery disease.
  Interventions: Combination Product: NVS Therapy

INTERVENTIONS:
Combination Product: NVS Therapy — Combination Product: NVS Therapy which includes NVS Injection (investigational product) and the following investigational devices: NVS Delivery Catheter, NVS Light Fiber, and NVS Light Source.
  Other Names: Natural Vascular Scaffold Therapy

SUMMARY:
The NVS Therapy is being studied to evaluate the safety and efficacy of retention of acute luminal gain, leading to acute hemodynamic improvement in superficial femoral and popliteal arteries with reference vessel diameters between 3.5 and 7.0 mm and lesion lengths between 36 and 96mm. The system is intended for use in patients with de novo lesions in the superficial femoral and proximal popliteal arteries.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center, open label Phase 1 study to assess the safety, pharmacokinetics (PK), and preliminary efficacy trends of applying NVS Therapy to de novo lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) during percutaneous transluminal angioplasty (PTA) in patients with life-style limiting claudication due to obstructive SFA and proximal popliteal artery atherosclerosis. Each investigator will receive supervised training for each procedure.

Eligibility to participate in the study is determined during the screening period and prior to the index procedure. Once a subject has been determined to be suitable for a peripheral intervention and all general eligibility criteria are met, angiographic eligibility will be evaluated at the time of the index procedure. Subjects then undergo the procedure with the NVS Therapy. Study data will be analyzed through the Day 365 follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject (or legal guardian) understands the study requirements and the treatment procedure and provides written informed consent before any study-specific tests or procedures are performed.
* Subject is eligible for PTA.
* Subject is willing to comply with all protocol required follow-up evaluations.
* Subject has documented Rutherford Classification 2 to 4 (see Appendix 3).
* Subject has laboratory test results that are within clinically acceptable limits.
* In Investigator's opinion, subject is hemodynamically stable at the time of the index procedure.
* Subject has a life expectancy of ≥1 year in the opinion of the Investigator.

Exclusion Criteria:

* Subject had cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 3 months prior to enrollment.
* Subject has any permanent neurologic defect that may cause non-compliance with the protocol.
* Subject had an MI within last the 3 months prior to enrollment.
* Subject is pregnant, planning to become pregnant, breastfeeding or planning to breastfeed in the next 365 days.
* Subject is currently receiving oral or intravenous immunosuppressive therapy (ie, inhaled steroids are not excluded).
* Subject has known life-limiting immunosuppressive or autoimmune disease (eg, human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus).
* Subject has local or systemic thrombolytic therapy within 48 hours prior to index procedure.
* Subject is currently on oral anticoagulation therapy, such as warfarin, rivaroxaban, apixaban, or dabigatran etexilate.
* Subject has known allergies or sensitivities to heparin, aspirin (ASA), or other anticoagulant/antiplatelet therapies.
* Subject has an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding.
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis.
* Subject has renal failure or chronic kidney disease with glomerular filtration rate (GFR) ≤ 30 mL/min or Modification of Diet in Renal Disease (MDRD) study equation result of ≤ 30 mL/min per 1.73 m2.
* Subject has white blood cell (WBC) count < (3,000 cells/mm3) within 7 days prior to index procedure.
* Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3 ≤ 7 days pre-procedure.
* Subject has been diagnosed with bleeding diatheses or hypercoagulable state.
* Subject has known or suspected active systemic infection evidenced by WBC > 14.0 (14,000/mm3).
* Subject is currently participating in another investigational drug or device study.
* Subject intends to participate in another investigational drug or device study within 365 days after the index procedure.
* Subject has any surgical procedure or intervention performed within the 30-day period prior to index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Freedom from all-cause mortality, target limb major amputation, and target lesion revascularization based on clinical observations | Day 30
  The overall composite occurrence of participants free from from all-cause mortality, target limb major amputation, and target lesion revascularization through post-index procedure to Day 30 will be summarized as a percentage.

OTHER OUTCOMES:
NVS Drug Plasma Concentrations | Day 1
  The Peak Plasma Concentration (Cmax) will be determined from plasma 10-8-10 Dimer concentrations for blood samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ansel, MD, Principal Investigator — OhioHealth Research Institute
Locations (3):
- United States (3):
  - OhioHealth Research Institute, Columbus, Ohio
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Wellmont CVA Heart Institute, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: No